CLINICAL TRIAL: NCT02908022
Title: Optimization of Brain-based Mechanisms Supporting Psychosocial Aspects of Acupuncture Therapy - a Hyperscanning fMRI Study
Brief Title: Brain Mechanisms of Psychosocial Aspects of Acupuncture Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Vitaly Napadow, Ph.D., Lic.Ac., Associate Professor, Harvard Medical School; Director, Center for Integrative Pain NeuroImaging (CiPNI), Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P002316; 4R33AT009306-03 (NIH)
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2024-10

CONDITIONS: Physician-patient Relationship; Fibromyalgia; Acupuncture Therapy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Interaction (Experimental): Phase 1:
  Prior to the MRI sessions, the clinician will be introduced to the patient and do a general intake of physical examination.
  During the MRI sessions, the patient will receive experimental pressure pain via the Hokanson Rapid Cuff Inflator and electroacupuncture analgesia to the leg for pain relief.
  Interventions: Device: Electroacupuncture Analgesia; Device: Hokanson Rapid Cuff Inflator
- No Interaction (Experimental): Phase 1:
  The clinician and the patient will first be introduced at the MRI sessions.
  During the MRI sessions, the patient will receive experimental pressure pain via the Hokanson Rapid Cuff Inflator and electroacupuncture analgesia to the leg for pain relief.
  Interventions: Device: Electroacupuncture Analgesia; Device: Hokanson Rapid Cuff Inflator
- Longitudinal (Experimental): Phase 2:
  Prior to first MRI session, both clinician and patient will go through a training visit.
  During the first MRI session, the patient will receive experimental pressure pain to the left leg via Hokanson Rapid Cuff Inflator and electroacupuncture to the same leg for pain relief.
  Following the first MRI session, the patient will attend biweekly acupuncture treatment sessions with the clinician (6 treatments total). During the first session the clinician will be introduced to the patient and do a general intake in addition to the acupuncture treatment.
  The final MRI session will be identical to the first. The patient will receive experimental pressure pain via Hokanson Rapid Cuff Inflator and electroacupuncture to the same leg for pain relief.
  Interventions: Device: Electroacupuncture Analgesia; Device: Hokanson Rapid Cuff Inflator

INTERVENTIONS:
Device: Electroacupuncture Analgesia — For the MRI sessions, acupuncture needles will be inserted next to the cuff placed on the left leg and will be connected to electrodes. Low-amplitude electrical current will be activated when a button is pressed via a handheld device, controlled by the acupuncturist, in order to reduce pain, acting as an analgesic.
  Additionally, electroacupuncture-induced analgesia will be used for the treatments. During the treatment sessions the acupuncturist will insert needles in several locations aimed to reduce the patient's fibromyalgia pain. Low-amplitude electrical current will be activated by the acupuncturist using the same electroacupuncture device as in the MRI machine.
Device: Hokanson Rapid Cuff Inflator — The Hokanson Rapid Cuff Inflator will be placed on the lower right leg of the subject and utilized for pain testing purposes according to the protocol. Ascending pressures will be administered using the cuff to elicit different pain intensities.

SUMMARY:
The overall aim of the present proposal is to investigate how patients' and clinicians' (Licensed acupuncturists, LAc) neural and autonomic processes during treatment interaction correlate to patient outcomes. Male and female healthy clinicians and fibromyalgia patients will be recruited for the study.

DETAILED DESCRIPTION:
First phase: At the training sessions, both clinician and patient will fill out a set of questionnaires and go through standardized psychophysical tests for assessing visual displays of affect. They will also be informed of the efficacy of the electroacupuncture in relieving pain during the experiment. During the clinical examination, the clinician will follow clinical exam protocol and do an intake of the fibromyalgia (FM) patient, including a physical exam and pain assessment. While in the scanner, the clinician will receive painful stimulations with a pressure cuff on the leg over an 8-minute paradigm in order to get cerebral representation. The patient will then be placed in a different scanner running simultaneously and will experience painful stimulations with a pressure cuff while interacting via live camera with the clinician in the other scanner. When visually prompted via cues on a screen, the clinician will activate analgesia for the patient, through a response device (response box) in clinician's one hand. After each trial of pain with/without treatment, the clinicians will be asked "how did you feel about the outcome (extremely positive - extremely negative)", and how satisfied are you (Not at all satisfied - Very satisfied) on Numerical Rating Scales (NRS). The patient will also give ratings after each trial of pain with/without treatment. They will be asked "how did you feel about the outcome (extremely positive - extremely negative)?", and "how painful was the cuff (Not painful - Extremely painful)?" on NRS. After the scan, both clinician and patient will be asked to rate anxiety during the presence of visual stimulus preceding cuff activation (not at all anxious - extremely anxious). After the final MRI session, the clinician and the patient will both be given the chance to report their responses to the treatment and then debriefed.

Second phase: At training session both clinician and patient will fill out a set of questionnaires. During the first MRI session the clinician will receive painful stimulations with a pressure cuff on the leg over a 6-minute paradigm in order to get cerebral representation. The patient will then be placed in a different scanner running simultaneously and will experience pain stimulation with the pressure cuff while interacting via live camera with the clinician in the other scanner. When visually prompted via cues on a screen, the clinician will activate analgesia for the patient, through a response device (response box) in clinician's hand. Both patient and acupuncturist will be asked to give ratings of pain and other parameters during the scan. Following the first MRI session, the patient will attend biweekly acupuncture treatment sessions with the clinician (6 treatments total). During the first session the clinician will be introduced to the patient and do a general intake in addition to the acupuncture treatment. The final MRI session will be identical to the first.

ELIGIBILITY:
Phase 1:

Inclusion Criteria (Healthy Clinicians):

* Male and Female healthy clinicians
* 25-60 years of age
* Ability to read and understand English; English can be a second language provided that the participant feels that he/she understand all the questions used in the assessment measures.

Inclusion Criteria (Fibromyalgia Patients):

* Have a clinical diagnosis of fibromyalgia and meet the Wolfe et al 2011 research criteria for fibromyalgia for at least one year
* Are on stable doses of medication for 30 days prior to entering the study and agree not to change medications or dosages during the trial
* 21 to 60 years of age
* Right-handed
* Ability to read and understand English; English can be a second language provided that the participant feels that he/she understand all the questions used in the assessment measures

Exclusion Criteria (All participants):

* Any longer period of work experience involving pain treatment, pain rehabilitation etc. This is in order to exclude participants with biased expectations regarding different methods of analgesia
* Presence of any illness or medication use that is judged to interfere with the trial. For example: psychiatric disorder according to the DSM-IV manual, medication that can influence cognition or emotional processing, i.e. sleep medication, antidepressants, anti-convulsants or opioids
* Presence of any contraindications to fMRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy
* Inability to respond accurately to the pain-relieving intervention in the behavioral part of the experiment, indicating a lack of response to the expectancy manipulation. If the healthy volunteer or clinician is not a responder to the behavioral expectancy induction he or she will be excluded
* Unwillingness to receive brief experimental pain
* Leg pain or health issues that may interfere with the study procedures

Exclusion Criteria (Specific to Fibromyalgia Patients):

* Comorbid acute pain condition
* Comorbid chronic pain condition that is rated by the subject as more painful than fibromyalgia
* Current use of opioid analgesics or stimulant medications or the fatigue associated with sleep apnea or shift work (e.g., modafinil)
* Documented peripheral neuropathy
* Any psychiatric disorder involving a history of psychosis (e. g schizophrenia, bipolar disorder, severe personality disorders)
* History of anxiety disorders or significant anxiety symptoms interfering with fMRI procedures (e.g., panic)
* Psychiatric hospitalization in the past 6 months
* Any impairment, activity or situation that in the judgment of the Study Coordinator or Principal Investigator would prevent satisfactory completion of the study protocol.
* Is an actual clinical patient of the clinician subject

Phase 2:

Inclusion Criteria (healthy individuals):

1. Male and female healthy clinicians.
2. 25-65 years of age (clinicians)
3. Ability to read and understand English; English can be a second language provided that the participant feels that he/she understand all the questions used in the assessment measures.

Inclusion Criteria (FM patients):

1. Have a clinical diagnosis of fibromyalgia and meet the Wolfe et al 2011 research criteria for fibromyalgia for at least one year
2. Are on stable doses of medication for 30 days prior to entering the study and agree not to change medications or dosages during the trial
3. 21-65 years of age
4. Ability to read and understand English; English can be a second language provided that the participant feels that he/she understand all the questions used in the assessment measures.

Exclusion Criteria (all participants):

1. Any longer period of work experience involving pain treatment, pain rehabilitation etc. This is in order to exclude participants with biased expectations regarding different methods of analgesia.
2. Presence of any illness that is judged to interfere with the trial. For example: psychiatric disorder according to the DSM-IV manual
3. Presence of any contraindications to fMRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy.
4. Inability to respond accurately to the pain-relieving intervention in the behavioral part of the experiment, indicating a lack of response to the expectancy manipulation. If the healthy volunteer or clinician is not a responder to the behavioral expectancy in-duction he or she will be excluded.
5. Unwillingness to receive brief experimental pain.
6. Leg pain or health issues that may interfere with the study procedures.

Exclusion Criteria (specific to FM patients):

1. Comorbid acute pain condition
2. Comorbid chronic pain condition that is rated by the subject as more painful than fibromyalgia
3. Documented peripheral neuropathy
4. Any psychiatric disorder involving a history of psychosis (e. g schizophrenia, bipolar disorder, severe personality disorders)
5. History of anxiety disorders or significant anxiety symptoms interfering with fMRI procedures (e.g., panic)
6. Psychiatric hospitalization in the past 6 months
7. Marijuana use greater than once daily and unwillingness to withhold from consumption 12 hours prior to scans or lab visits
8. Unwillingness to withhold from consuming nicotine 4 hours prior to scans
9. Any impairment, activity or situation that in the judgment of the Study Coordinator or Principal Investigator would prevent satisfactory completion of the study protocol.
10. Is an actual clinical patient of the clinician subject

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-09; Primary Completion 2024-05 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
Magnitude of patient/clinician concordance in brain activation of mirror brain circuitry during electroacupuncture therapy | Up to 60 months
  Patient/clinician concordance in brain activation will be assessed by functional Magnetic Resonance Imaging, simultaneously for both the patient and the clinician

SECONDARY OUTCOMES:
Correlation between patient/clinician brain activity concordance and pain relief from electroacupuncture therapy | Up to 60 months
  Patient/clinician concordance in brain activation will be assessed by functional Magnetic Resonance Imaging, simultaneously for both the patient and the clinician

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Napadow, PhD, LicAc, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (2):
- United States (2):
  - Martinos Center for Biomedical Imaging, Charlestown, Massachusetts
  - Spaulding Rehabilitation Hospital, Charlestown, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schliessbach J, van der Klift E, Arendt-Nielsen L, Curatolo M, Streitberger K. The effect of brief electrical and manual acupuncture stimulation on mechanical experimental pain. Pain Med. 2011 Feb;12(2):268-75. doi: 10.1111/j.1526-4637.2010.01051.x. Epub 2011 Jan 28. PMID 21276188
- [Background] Lang PM, Stoer J, Schober GM, Audette JF, Irnich D. Bilateral acupuncture analgesia observed by quantitative sensory testing in healthy volunteers. Anesth Analg. 2010 May 1;110(5):1448-56. doi: 10.1213/ANE.0b013e3181d3e7ef. Epub 2010 Mar 17. PMID 20237044
- [Background] Zheng Z, Feng SJ, Costa Cd, Li CG, Lu D, Xue CC. Acupuncture analgesia for temporal summation of experimental pain: a randomised controlled study. Eur J Pain. 2010 Aug;14(7):725-31. doi: 10.1016/j.ejpain.2009.11.006. Epub 2009 Dec 31. PMID 20045360
- [Background] Cruz-Almeida Y, Fillingim RB. Can quantitative sensory testing move us closer to mechanism-based pain management? Pain Med. 2014 Jan;15(1):61-72. doi: 10.1111/pme.12230. Epub 2013 Sep 6. PMID 24010588
- [Background] Naeser MA, Hahn KA, Lieberman BE, Branco KF. Carpal tunnel syndrome pain treated with low-level laser and microamperes transcutaneous electric nerve stimulation: A controlled study. Arch Phys Med Rehabil. 2002 Jul;83(7):978-88. doi: 10.1053/apmr.2002.33096. PMID 12098159
- [Background] Gabriel A, Sobota R, Gialich S, Maxwell GP. The use of Targeted MicroCurrent Therapy in postoperative pain management. Plast Surg Nurs. 2013 Jan-Mar;33(1):6-8; quiz 9-10. doi: 10.1097/PSN.0b013e3182844219. PMID 23446501
- [Background] Gossrau G, Wahner M, Kuschke M, Konrad B, Reichmann H, Wiedemann B, Sabatowski R. Microcurrent transcutaneous electric nerve stimulation in painful diabetic neuropathy: a randomized placebo-controlled study. Pain Med. 2011 Jun;12(6):953-60. doi: 10.1111/j.1526-4637.2011.01140.x. Epub 2011 May 31. PMID 21627767